CLINICAL TRIAL: NCT05512390
Title: A First In Human Multicenter, Open-Label Study to Determine the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ABBV-319 in B-cell Malignancies
Brief Title: A Study to Assess the Adverse Events, Change in Disease Activity, and How Intravenously Infused ABBV-319 Moves Through the Bodies of Adult Participants With Relapsed or Refractory (R/R) Diffuse Large B-cell Lymphoma (DLBCL), Follicular Lymphoma (FL), or Chronic Lymphocytic Leukemia (CLL)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M22-716
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B-Cell Lymphoma; Chronic Lymphocytic Leukemia; Follicular Lymphoma
Keywords: Diffuse Large B-Cell Lymphoma; Chronic Lymphocytic Leukemia; Follicular Lymphoma; Cancer; B-Cell Malignancies; ABBV-319
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose Escalation ABBV-319 (Experimental): Participants with relapsed or refractory (R/R) B cell lymphomas including diffuse large b-cell lymphoma (DLBCL) or follicular lymphoma (FL), and Chronic lymphocytic leukemia (CLL) will receive escalating doses of ABBV-319 in 21-day cycles, until the doses of ABBV-319 that will be used in the next phase are determined.
  Interventions: Drug: ABBV-319
- (ABBV-319) Diffuse Large B-cell Lymphoma (DLBCL) Participants (Experimental): Participants with R/R DLBCL will receive ABBV-319 in 21-day cycles.
  Interventions: Drug: ABBV-319
- (ABBV-319) Follicular Lymphoma (FL) Participants (Experimental): Participants with R/R FL will receive ABBV-319 in 21-day cycles.
  Interventions: Drug: ABBV-319
- (ABBV-319) Chronic Lymphocytic Leukemia (CLL) Participants (Experimental): Participants with R/R CLL will receive ABBV-319 in 21-day cycles.
  Interventions: Drug: ABBV-319

INTERVENTIONS:
Drug: ABBV-319 — Intravenous (IV); Infusion

SUMMARY:
B-cell Lymphoma is an aggressive and rare cancer of a type of immune cells (a white blood cell responsible for fighting infections). Follicular Lymphoma is a slow-growing type of non-Hodgkin lymphoma. Chronic lymphocytic leukemia (CLL) is the most common leukemia (cancer of blood cells). The purpose of this study is to assess the safety, tolerability, pharmacokinetics, and preliminary efficacy of ABBV-319 in adult participants in relapsed or refractory (R/R) diffuse large b-cell lymphoma (DLBCL), R/R follicular lymphoma (FL), or R/R CLL. Adverse events will be assessed.

ABBV-319 is an investigational drug being developed for the treatment of R/R DLBCL, R/R FL, or R/R CLL. This study will include a dose escalation phase to determine the doses of ABBV-319 that will be used in the next phase and a dose expansion phase to determine the change in disease activity in participants with R/R DLBCL, R/R FL, and R/R CLL. Approximately 154 adult participants with R/R B cell lymphomas including R/R DLBCL, R/R FL, and R/R CLL will be enrolled in the study in sites world wide.

In the Dose Escalation phase of the study participants will receive escalating intravenously infused doses of ABBV-319 in 21-day cycles, until the Phase 2 dose is determined. In the dose expansion phase of the study participants receive intravenously infused ABBV-319 in 21-day cycles.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* For dose escalation (Part 1) only: Participants with documented diagnosis of B-cell malignancies including those with histology based on criteria established by the World Health Organization (WHO), and measurable disease requiring treatment, as per the protocol.
* For the relapsed or refractory diffuse large b-cell lymphoma (DLBCL), follicular lymphoma (FL), and Chronic lymphocytic leukemia (CLL) dose expansion cohorts (Part 2) only: Participants with documented diagnosis of one of the B-cell malignancies noted in the protocol with histology based on criteria established by the WHO, and measurable disease requiring treatment, as per the protocol.
* Laboratory values meeting the criteria noted in the protocol.
* For participants previously treated with a CD19-targeting therapy (eg, CD19 monoclonal antibody) a core or excision tumor biopsy subsequent to the most recent CD19-targeting therapy must be collected.
* Participant must have measurable disease, as defined by the 2014 Lugano Classification.

Exclusion Criteria:

* Known active central nervous system (CNS) disease, or primary CNS lymphoma.
* Known active infection or clinically significant uncontrolled conditions as per the protocol.
* Eastern Cooperative Oncology Group (ECOG) performance status >= 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of Dose-Limiting Toxicities (DLT) | Day 42
  A DLT is defined as any adverse event (AE) for which a clear alternative cause cannot be established (eg, attributed to the disease under study, another disease, or to a concomitant medication by the study investigators or medical monitor).
Number of Participants with Adverse Events (AE) | Up to 30 Months
  AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Maximum Observed Serum Concentration (Cmax) of ABBV-319 | Up to 6 Months
  Maximum observed serum concentration of ABBV-319.
Time to Cmax (Tmax) of ABBV-319 | Up to 6 Months
  Time to Cmax of ABBV-319.
Terminal Phase Elimination Half-Life (t1/2) of ABBV-319 | Up to 6 Months
  Terminal phase elimination half-life of ABBV-319.
Area Under the Serum Concentration Versus Time Curve (AUC) of ABBV-319 | Up to 6 Months
  Area under the serum concentration versus time curve (AUC) of ABBV-319.
Antidrug Antibody (ADA) | Up to 6 Months
  Incidence and concentration of anti-drug antibodies.

SECONDARY OUTCOMES:
Number of Participants with Response of Partial Response (PR) or Better per Disease-Specific Criteria | Up to 6 Months
  Number of participants with response of PR or better per disease-specific criteria.
Duration of Response (DOR) | Up to 6 Months
  DOR is defined for participants achieving a complete response (CR)/PR as the time from the initial response per investigator review to disease progression or death of any cause, whichever occurs earlier.
Time to Response | Up to 6 Months
  Time to response is defined for participants achieving a CR/PR as the time from starting therapy to first a CR/PR.
Progression Free Survival (PFS) Time | Up to 30 Months
  PFS is defined as time from first study treatment to a documented disease progression as determined by the investigator, or death due to any cause, whichever occurs earlier.
Overall survival (OS) Time | Up to 30 Months
  OS is defined as time from first study treatment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (20):
- United States (8):
  - University of Arizona Cancer Center - Tucson /ID# 247752, Tucson, Arizona
  - Sylvester Comprehensive Cancer Center - University of Miami /ID# 247232, Miami, Florida
  - Allina Health System /ID# 251782, Minneapolis, Minnesota
  - University of Nebraska Medical Center /ID# 246715, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 249246, New York, New York
  - Novant Health Presbyterian Medical Center /ID# 246719, Charlotte, North Carolina
  - Baylor Sammons Cancer Center /ID# 247715, Dallas, Texas
  - University of Texas Health San Antonio MD Anderson Cancer Center /ID# 256234, San Antonio, Texas
- Australia (3):
  - Concord Repatriation General Hospital /ID# 249240, Concord, New South Wales
  - St Vincent's Hospital Melbourne /ID# 247624, Fitzroy Melbourne, Victoria
  - One Clinical Research Pty Ltd /ID# 248392, Nedlands, Western Australia
- Canada (2):
  - Cross Cancer Institute /ID# 246717, Edmonton, Alberta
  - University Health Network_Princess Margaret Cancer Centre /ID# 243936, Toronto, Ontario
- Israel (2):
  - The Chaim Sheba Medical Center /ID# 254884, Ramat Gan, Tel Aviv
  - Hadassah Medical Center-Hebrew University /ID# 254885, Jerusalem
- South Korea (3):
  - Seoul National University Hospital /ID# 263945, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 263220, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 263294, Seoul, Seoul Teugbyeolsi
- Spain (2):
  - Hospital Universitario Marques de Valdecilla /ID# 262826, Santander, Cantabria
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 265198, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-716